CLINICAL TRIAL: NCT06071819
Title: Generalized Anxiety Disorder and Panic Disorder: Differences in Clinical Manifestation and Prognosis, a Multicenter Study
Brief Title: Clinical Markers of Panic and Generalized Anxiety Disorder
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Alice Caldiroli, Psychiatrist, University of Milano Bicocca
Other Study IDs: GAD-PD-3955
Record Dates: First submitted 2023-01-05; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder; Duration of Untreated Illness
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Generalized Anxiety Disorder (GAD): Patients affected by GAD
  Interventions: Diagnostic Test: Structured Clinical Interview for DSM-5
- Panic Disorder (PD): Patients affected by Panic Disorder
  Interventions: Diagnostic Test: Structured Clinical Interview for DSM-5

INTERVENTIONS:
Diagnostic Test: Structured Clinical Interview for DSM-5 — A structured interview will be administered to confirm the diagnosis reported in clinical charts

SUMMARY:
The goal of this observational study is to compare socio-demographic and clinical features in patients affected by Generalized Anxiety Disorder (GAD) and by Panic Disorder (PD). The main questions it aims to answer are:

* which socio-demographic/clinical markers are associated to GAD or PD diagnosis?
* which factors are associated with a longer duration of untreated illness (DUI) in GAD and in PD? Participants will signed a written informed consent and socio-demographic/clinical variables will be retrospectively collected. Researchers will compare GAD and PD groups in terms of socio-demographic and clinical features, including DUI, to better characterize the two disorders and to investigate factors associated to a longer DUI.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years;
* ability and willing to give informed consent;
* fluency in Italian language;
* diagnosis of GAD or PD according to the criteria of the Diagnostic and Statistical Manual of Mental Disorder, 5th edition.

Exclusion Criteria:

* intellectual disability;
* lack of clinical and socio-demographic information;
* patients treated for less than three months in the outpatient clinics for the impossibility of a comprehensive collection of clinical variables.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients suffering from PD or GAD identified from medical records in the pre-pandemic period (2016-2019).
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Quantitative socio-demographic / clinical variables | Three months
  Age (years), age at onset (years), duration of illness (years), duration of treatment (years)
Sex | Three months
  Sex (male/female)
Occupation | Three months
  Occupation (employed/unemployed)
Pre-/post-onset Comorbidity | Three months
  Psychiatric and medical comorbidity
Substance misuse | Three months
  Substance misuse
Treatment | Three months
  Treatment, treatment discontinuation and side effects
Dichotomous socio-demographic / clinical variables | Three months
  Multiple family history of psychiatric disorders (yes/no), pre- and post-onset psychiatric poly-comorbidities (yes/no), presence of personality disorder (yes/no), pre- and post-onset poly-substance misuse (yes/no), pre- and post-onset medical poly-comorbidities (yes/no), suicide attempts (yes/no), hospitalizations (yes/no), poly-therapy (yes/no), presence of poly-side effects (yes/no), presence of lifetime psychotherapy (yes/no)

SECONDARY OUTCOMES:
Duration of untreated illness (DUI) in months = time between the onset of PD and the first appropriate pharmacological treatment. | Three months
  Factors associated to DUI among GAD and PD groups. Information about DUI have been registered according to what the patient reported (clinical records and structured interviews)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Caldiroli, Doctor, Principal Investigator — University of Milano Bicocca - Fondazione IRCCS San Gerardo dei Tintori
Locations (1):
- University of Milano Bicocca - Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided